CLINICAL TRIAL: NCT01569724
Title: Estimation of Carbohydrate Metabolism Disorder Frequency in Hypertriglyceridemia Induced by Bexarotene Treatment of Cutaneous T Cell Lymphoma - Pilote Study
Brief Title: Carbohydrate Metabolism Disorder Frequency in Hypertriglyceridemia Induced by Bexarotene of Cutaneous T Cell Lymphoma
Acronym: TgBEX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-A23465-21
Record Dates: First submitted 2012-02-24; First posted 2012-04-03 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Hypertriglyceridemia; Cutaneous T Cell Lymphoma
Keywords: hypertriglyceridemia; bexarotene
MeSH Terms: conditions — Hypertriglyceridemia; Lymphoma, T-Cell, Cutaneous | interventions — Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- bexarotene (Experimental)
  Interventions: Other: oral glucose tolerance test (OGTT)

INTERVENTIONS:
Other: oral glucose tolerance test (OGTT) — patients presenting an hypertriglyceridemia will have a oral glucose tolerance test (OGTT) in order to diagnose a carbohydrate metabolism disorder
  Other Names: Non applicable.

SUMMARY:
Bexarotene is a RXR-selective retinoid, licensed for the treatment of cutaneous T cell lymphoma. The most frequent adverse effect is hypertriglyceridemia but its mechanism is not well known. The purpose of this study is to research a carbohydrate metabolism disorder associated in bexarotene-induced hypertriglyceridemia.

DETAILED DESCRIPTION:
Primary cutaneous lymphomas are the second group of extra nodal lymphomas after gastrointestinal lymphomas. Bexarotene is licensed for the treatment of epidermotropic cutaneous T cell lymphoma .The most common side effect of bexarotene is hypertriglyceridemia (82%) associated with hypercholesterolemia (30 to 40%). Central hypothyroidism is also present in 40-80% of cases. These adverse effects are dose-dependent. The management of hyperlipidemia induced by bexarotene is difficult. The mechanism of lipid disorder induced by bexarotene is not well known. Associated carbohydrate metabolism disorder could be present and play a role in the bexarotene-induced hyperlipidemia.

The main objective is to estimate the frequency of a carbohydrate disorder in patients with hypertriglyceridemia (TG> 1.5 g / L) induced by bexarotene treatment of cutaneous T cell lymphoma, previously free of diabetes, thyroid dysfunction and dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18 years
* Diagnosis of epidermotropic CTCL confirmed by histological examination for which consideration will be given treatment with bexarotene due to the advanced stage of lymphoma (stage IIB-IV) or earlier stage if resistance to previous treatment .
* TSH, FT3 and FT4 within normal limits
* AST and ALT ≤ 2 * upper limit of normal
* Creatinine clearance ≥ 30 mL / min
* Agreement after written information and informed to participate in the study
* Patient accepting the constraints of the study
* Membership of a social security system.

Exclusion Criteria:

* Pregnant or lactating woman
* Women of childbearing potential without effective contraception
* Insufficient thyroid or hyperthyroidism
* Diabetes known or detected
* Hyperlipidemia known or detected
* Hepatic insufficiency
* Difficulties to understand
* Persons covered by a plan of legal protection (protection of justice, guardianship, curator) or unable to issue a consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-01; Primary Completion 2016-12 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
glucose intolerance or diabetes | At 0, 2, 4, 6, 8 weeks after the administration of bexarotene.
  The presence of a carbohydrate disorder is defined by glucose intolerance or diabetes. The diagnosis of glucose intolerance is made for a fasting glucose less than 1.26 g / l glucose and 2 hours (T120mn) after taking 75 g of glucose during an oral glucose tolerance test (OGTT) between 1.4 and 2 g / l and / or a value greater than or equal to 2 g / l between T30 and T90 min. Diabetes is established for a fasting glucose greater than or equal to 1.26 g / l and / or blood glucose greater than or equal to 2 g / l to 2 hours.

SECONDARY OUTCOMES:
hypothyroidism | At 0, 2, 4, 6, 8 weeks after the administration of bexarotene.
  hypothyroidism detection: TSH, free T3 and free T4 measured weekly during the first month and then every 15 days in the second month. Laboratory abnormalities will be evaluated according to the standards of the laboratory of each center.
response to bexarotene | At 0, 2, 4, 6, 8 weeks after the administration of bexarotene.
  Response to bexarotene: it is considered partial if the patient has a decrease in injuries between 50% and 90% to total as if it has a lower damage of more than 90%.

CONTACTS AND LOCATIONS:
Overall Officials: Henri ADAMSKI, MD, Principal Investigator — Rennes University Hospital; Emmanuel OGER, MD, PhD, Study Chair — Rennes University Hospital
Locations (1):
- Service de dermatologie - Hôpital de Pontchaillou, Rennes, France